CLINICAL TRIAL: NCT03091426
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Pharmacodynamics, Safety, Tolerability and Efficacy of Omiganan BID in Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Pharmacodynamics of Omiganan BID in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-014; 2016-003849-28 (EudraCT Number)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Omiganan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Omiganan 1% (Experimental)
  Interventions: Drug: Omiganan
- Omiganan 1.75% (Experimental)
  Interventions: Drug: Omiganan
- Omiganan 2.5% (Experimental)
  Interventions: Drug: Omiganan
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omiganan — Omiganan 1%
  Arms: Omiganan 1%
Drug: Omiganan — Omiganan 1.75%
  Arms: Omiganan 1.75%
Drug: Omiganan — Omiganan 2.5%
  Arms: Omiganan 2.5%
Drug: Placebo — Vehicle
  Arms: Vehicle

SUMMARY:
This study has a randomized, double-blind, placebo-controlled design to assess the efficacy, pharmacodynamics and safety/tolerability of omiganan in patients with mild to moderate atopic dermatitis when applied BID to all atopic dermatitis lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with mild to moderate AD (IGA 2 or 3) 18 to 65 years of age,inclusive. The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease other than AD following a detailed medical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, virology and urinalysis;
* Confirmed AD diagnosis;
* Symptoms present for at least 1 year;
* EASI between 7.1 - 50.0, inclusive at screening;
* 2-20% body surface area (BSA) affected at screening;
* Body mass index (BMI) between 18 and 35 kg/m2, inclusive, and with a minimum weight of 50 kg;
* Able to participate and willing to give written informed consent and to comply with the study restrictions;
* Subjects and their partners of childbearing potential must use effective contraception, for the duration of the study and for 3 months after the last dose.

Exclusion Criteria:

* Any current and / or recurrent clinical significant skin condition other than AD;
* Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding;
* Ongoing use of prohibited atopic dermatitis treatments. Requires washout period prior to baseline (first dose of the study drug);
* Use of topical medication (prescription or over-the-counter [OTC]) within 14 days of study drug administration, or less than 5 half-lives (whichever is longer) in local treatment area;
* Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment;
* Known hypersensitivity to the compound or excipients of the compound or known hypersensitivity to one or more different emollients;
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year;
* Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation (oSCORAD) | Within 7 Weeks
  oSCORAD Assessment
Clinical Evaluation (EASI) | Within 7 Weeks
  EASI Assessment
Clinical Evaluation (IGA) | Within 7 Weeks
  IGA Assessment
Patient-Orientated Outcome Measure (POEM) | Within 7 Weeks
  Patient Assessment by collecting POEM
Dermatology Life Quality Index (DLQI) | Within 7 Weeks
  Assessment of health-related quality of life by measuring DLQI
eDiary | Within 4 Weeks
  Singe-Question assessment of pruritus and sleeplessness
Clinical Photography | Within 7 Weeks
  Whole body photograph for qualitative and observational record
Pharmacodynamics (Biomarkers) | Within 7 Weeks
  Local biomarkers sequencing
Pharmacodynamics (Microbiome) | Within 7 Weeks
  Microbiome analysis
Pharmacodynamics (Microbiology) | Within 7 Weeks
  Microbiology analysis
Pharmacodynamics (TEWL) | Within 7 Weeks
  Transepidermal water-loss assessment
Pharmacodynamics (Thermography) | Within 7 Weeks
  Skin temperature measurements will be taken
Pharmacodynamics (TAP) | Within 7 Weeks
  Analysis of biomarkers captured by Transdermal Analysis Patch
Pharmacodynamics (Cytokines) | Within 7 Weeks
  Cytokine assessment via blood evaluation

SECONDARY OUTCOMES:
Safety (AE) | Within 7 Weeks
  Adverse Events will be collected throughout the study
Safety (Vital Signs) | Within 7 Weeks
  Vital Signs will be collected throughout the study
Safety (Clinical Laboratory Tests) | Within 7 Weeks
  Lab samples collected in various timepoints within the study
Safety (ECG) | Within 7 Weeks
  ECGs collected before beginning and end of study

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- LUMC/Centre for Human Drug Research, Leiden, Netherlands